CLINICAL TRIAL: NCT00438308
Title: Prospective Randomized Comparison of Early and Late Wrist Mobilization After Volar Plate Fixation of a Fracture of the Distal Radius
Brief Title: Comparison of Early and Late Therapy for Adults With Operatively Treated Distal Radius Fractures
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: David C Ring, MD, Massachusetts General Hospital
Other Study IDs: 2004-P-002118
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Distal Radius Fractures
Keywords: distal radius fracture; rehabilitation; volar plate fixation; DASH questionnaire
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Subjects who begin therapy immediately after fracture.
- 2: Subjects delay therapy for 3 weeks after injury.

SUMMARY:
The purpose of the study is to compare two common ways of rehabilitating after surgery for distal radius fractures treated operatively with a volar plate.

DETAILED DESCRIPTION:
Over the last three decades, operative treatment of distal radius fractures has become increasingly common compared to non-operative treatment. Over the last 15 years there has been a trend towards more invasive, internal plate fixation of fractures of the distal radius. One argument in favor of internal fixation for these fractures is that, similar to other periarticular fractures, it would be beneficial to allow early movement of the wrist articulation. There is not, however, any data to support this statement. In fact, data regarding external fixation that either immobilizes the wrist or allows wrist motion suggest that early wrist mobilization is not as important as the overall alignment of the bone in terms of final wrist motion. This question is important in patient care and in decision-making regarding these fractures. Additionally, many companies use this claim as a marketing point in spite of the lack of evidence. We consider that good quality data is needed to determine the answer to this issue and to help to resolve the related problems described above.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or female
* Age: Older than 18
* Isolated distal radial fracture
* Fracture treated with volar plates, stable fixation
* Initial treatment within 4 weeks of trauma

Exclusion Criteria:

* Complex fractures that require additional or different material than volar plates
* Unstable fractures in which early mobilization is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the MGH Hand and Upper Extremith Service
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2004-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
range of motion in degrees of the wrists | 6 months

SECONDARY OUTCOMES:
DASH score | 6 months
Likert pain scale | 6 months
pinch and grip strength | 6 months
Gartland and Werely score | 6 months
and Mayo wrist score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital